CLINICAL TRIAL: NCT02975648
Title: Effect of an Educational Model on Physical Activity in Individuals Undergoing the First Percutaneous Coronary Intervention: Randomized Clinical Trial
Brief Title: Educational Model for Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Natássia Condilo Pitta, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 51805715.0.0000.5393
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease; Coronary Disease; Arteriosclerosis; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Arteriosclerosis; Cardiovascular Diseases | interventions — Models, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): At discharge, paticipants received guidance from health professionals. The paticipants had a medical return five to seven months after the percutaneous coronary intervention.
  Interventions: Behavioral: usual care
- Educational model + follow up (Experimental): The paticipants received the hospital's instructions at discharge and participated in the educational program (booklets with telephone follow-up). The paticipants had a medical return five to seven months after discharge
  Interventions: Behavioral: educational model + follow up

INTERVENTIONS:
Behavioral: educational model + follow up — Orientation from health professionals at discharge, educational program with explanation of booklets and telephone follow-up (three calls)
  Arms: Educational model + follow up
Behavioral: usual care — Hospital health professionals offered orientation on care after discharge
  Arms: Usual Care

SUMMARY:
The purpose of this study was to compare the effect of an educational model, which included cardiac rehabilitation with emphasis on physical activity and telephone follow up, with the usual management of individuals undergoing to first percutaneous coronary intervention, in relation to physical activity five until seven months after discharge.

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) at a public teaching hospital, which has specialized care for CAD in Ribeirão Preto, state of São Paulo, Brazil. The intervention group received usual care and an educational programme and the control group received only usual care.

A researcher (who didn't had contact with the patients) generated the random allocation in SPSS software, concealing it from the investigators in sequentially numbered, sealed and opaque envelopes.

Another researcher performed the individual interview with each participant (baseline) and aplied the instruments of socialdemographic data, physical activity, ansiety and depression, perceived health status and selfefficacy to practice of physical activity. At the end of the interviewThe same researcher opened the envelope to allocate the participants to either intervention or control group. The participants of intervention group remained with the researcher to receive the intervention.

The educational programme consisted of four booklets entitled 1. Percutaneous Transluminal Coronary Angioplasty, 2. Going home after your coronary angioplasty, 3. How to take care of your heart and your health, and 4. How to practice physical activities. The educational programme included the telephone follow-up that contained three calls to motivate the participants to change their lifestyle and clarify doubts. The contents of the booklets were explained step by step to the participants by the researcher who conducted the interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or more) of both genders
* Patients undergoing the first percutaneous coronary intervention
* Patients who had a properly functioning home phone line

Exclusion Criteria:

* No cognitive conditions to participate (assessed by the ability to inform the name, current date, day of the week, place, age and place of birth confirmed by the participant's identification document)
* Who did not have clinical or physical conditions to answer the questionnaires (individuals with dyspnea and / or mental confusion)
* Who reported difficulties to speak on the phone (hearing loss)
* Who had sequelae that could influence activities of daily living (limb amputation or paralysis)
* Who had a contraindication to physical exercise, prescribed by the doctor, and who already participated in a supervised cardiac rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in physical activity level from baseline to five to seven months | baseline and five to seven months
  The "Baecke Questionnaire of Habitual Physical Activity" was developed by Baecke, Burema and Frijters (1982) and validated for the Brazilian population by Florindo et al. (2004, 2006). The instrument has three dimensions: occupational physical activity (eight questions), physical activity during leisure time (four questions) and leisure and locomotion activities (four questions), totaling 16 questions. Higher scores indicate a higher level of physical activity. This questionnaire was used to collect the data at baseline and five to seven months after hospital discharge.

SECONDARY OUTCOMES:
Change in symptoms of anxiety and depression from baseline to five to seven months | baseline and five to seven months
  The questionnaire "Hospital Anxiety and Depression Scale" was developed by Zigmond and Snaith (1983) and validated and adapted to Portuguese by Botega et al. (1995). The Hospital Anxiety and Depression Scale contains 14 multiple choice questions, divided into two subscales: anxiety and depression (composed of seven items each). Higher scores indicate more symptoms of anxiety and depression. This questionnaire was used to collect the data at baseline and five to seven months after hospital discharge.
Change in perceived health status from baseline to five to seven months | baseline and five to seven months
  The questionnaire "Medical Outcomes Survey 36 - Item Short-Form" developed by Ware and Sherboune (1992). The investigators used the version licensed by Quality Metric Incorporated (MARUISH, 2011) for use in surveys in Brazil. The Medical Outcomes Survey 36 - Item Short-Form is a multidimensional questionnaire composed of 36 items that evaluate eight health concepts: functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects, mental health and a comparative question that evaluate the current health conditions with one year ago. Higher values indicate better perceived health status. This questionnaire was used to collect the data at baseline and five to seven months after hospital discharge.
Change in self-efficacy for physical activity from baseline to five to seven months | baseline and five to seven months
  The questionnaire "Escala de Autoeficácia Para Prática de Atividade Física" developed by Rech et al. (2011) for Brazilian adults and by Borges et al. (2015) that used in the elderly population. This questionnaire was elaborated from two specific scales of self-efficacy for the practice of physical exercise, proposed by Sallis et al. (1988) and Bandura (2006). We used the Brazilian adult version (RECH et al., 2011) which contains two domains with five items each in which the answers are dichotomous ( "no" versus "yes"). Higher scores indicate better self-efficacy for physical activity. The instrument was used to collect the data at baseline and five to seven months after hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia A Rossi, PhD, Study Chair — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No